CLINICAL TRIAL: NCT02416960
Title: Effect of a Hypocaloric Diet With Different Glycemic Indexes on Ghrelin and Leptin Levels, Metabolic Parameters, and Reproductive Outcomes in Overweight and Obese Infertile Women: A Randomized Clinical Trial
Brief Title: Effect of the Glycemic Index of Diet on Metabolic and Reproductive Parameters in Overweight and Obese Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11-0326
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Female Infertility; Obesity
Keywords: female infertility; glycemic index; leptin; ghrelin; overweight; obesity; in vitro fertilization
MeSH Terms: conditions — Infertility, Female; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Glycemic Index Diet Group (Experimental): Patients will follow a treatment with a hypocaloric diet with low glycemic index/load for 12 weeks, immediately before the in vitro fertilization cycle.
  Interventions: Other: Low Glycemic Index Diet Group
- Conventional Diet Group (Active Comparator): Patients will follow a treatment with a hypocaloric diet with high glycemic index/load for 12 weeks, immediately before the in vitro fertilization cycle.
  Interventions: Other: Conventional Diet Group
- Control Group (No Intervention): Patients will follow their usual diet for 12 weeks, immediately before the in vitro fertilization cycle.

INTERVENTIONS:
Other: Low Glycemic Index Diet Group — This diet will be designed as a moderate reduced-energy, moderate-to-high ﬁber, low glycemic index/load diet.
  Arms: Low Glycemic Index Diet Group
Other: Conventional Diet Group — This diet will be designed as a moderate reduced-energy, moderate-to-high ﬁber, high glycemic index/load diet.
  Arms: Conventional Diet Group

SUMMARY:
Infertility has been currently recognized as a disorder related to obesity. Among several metabolic changes associated with obesity, insulin resistance appears to be linked to hormonal disorders that affect reproductive system. Leptin and ghrelin are hormones involved in energy balance regulation and are also associated with reproductive system regulation, but its relationship with infertility is scarce. The aim of this study is to determine the effect of a hypocaloric diet with different glycemic indexes on ghrelin and leptin levels, hormonal, metabolic and reproductive parameters in infertile overweight or obese women candidates to in vitro fertilization. The patients who meet the inclusion criteria and accept to participate in the study, will be allocated in one of the following groups: Hypocaloric Low Glycemic Index diet group; Hypocaloric Conventional diet group or Control group (maintenance of usual diet) and follow the study protocol for 12 week. Immediately after the end of the diet protocol, the patients will be submitted to the in vitro fertilization treatment.

DETAILED DESCRIPTION:
Infertility has been currently recognized as a disorder related to obesity. Among several metabolic changes associated with obesity, insulin resistance appears to be linked to hormonal disorders that affect reproductive system. Leptin and ghrelin are hormones involved in energy balance regulation and are also associated with reproductive system regulation, but its relationship with infertility is scarce. The aim of this study is to determine the effect of a hypocaloric diet with different glycemic indexes on ghrelin and leptin levels, hormonal, metabolic and reproductive parameters in infertile overweight or obese women candidates to in vitro fertilization. Infertile women with grade I and II obesity, or pre-obesity with increased waist circumference will be recruited. Patients will be assigned to Hypocaloric Low Glycemic Index diet group; Hypocaloric Conventional diet group or Control group (maintenance of usual diet), and will follow the protocol for 12 weeks. The two intervention diets will be similar in terms of caloric intake and macronutrient distribution and different in terms of carbohydrates quality (index and glycemic load). Immediately after the end of the diet protocol, the patients will be submitted to the in vitro fertilization treatment. Before and after the intervention anthropometric measurements (weight, height, body mass index, waist and hip circumference) and body composition (body fat percentage determined by the measurement of seven skinfolds) will be evaluated as well as biochemical parameters: leptin, acylated ghrelin, glucose, insulin, serum lipids (total cholesterol and lipoproteins, and triglycerides), sex hormones - follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol, progesterone, prolactin, testosterone and sex hormone binding globulin (SHBG). Primary outcome: clinical pregnancy rate. Secondary outcomes: HOMA-IR (Homeostasis Model Assessment), acylated ghrelin and leptin levels, body fat percentage, number of oocytes retrieved, percentage of fertilized oocytes and embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of female infertility and indication for treatment with in vitro fertilization
* Body Mass Index (BMI) equal or greater than 30 kg/m² or BMI > 25 kg/m² with increased waist circumference (> 80 cm);
* Being not treated (diet) for weight loss/gain and maintaining stable body weight in the three months prior to the study;
* Not having stomach/digestive problems
* Not having the knowledge of cardiovascular disease history;
* Non-smokers;
* Not using any medication.

Exclusion Criteria:

* Patients with BMI equal or higher than 40 kg/m² (morbid obesity)
* Patients who are already receiving some type of nutritional intervention
* Patients with co-morbidities that may interfere with reproductive capacity (genetic and/or endocrine disorders, diabetes mellitus, cancer, liver or kidney failure), alcoholics, individuals who have contact (work) with heavy metals or chemicals (exposure to solvents and pesticides)
* Lack of adherence to the proposed dietary treatment

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | up to 18 weeks - in average, two weeks after the end of the in vitro fertilization cycle
  Clinical Pregnancy will be considered as pregnancy diagnosed by ultrasound visualization of one or more gestational sacs or definitive clinical signs of pregnancy.

SECONDARY OUTCOMES:
HOMA-IR index (Homeostasis Model Assessment) | baseline and 12 weeks
  The HOMA-IR index will be obtained by the following formula: fasting glucose (mg/dl/18) x fasting insulin (U/mL)/22.5.
Acylated Ghrelin Levels (pg/dL) | baseline and 12 weeks
  The levels of acylated ghrelin will be determined by enzyme immunoassay (SPI BIO, Montigny le Bretonneux, France) using a plate reader (Biochrom Anthos MultiRead 400, Biochrom Ltd., Cambridge, UK).
Leptin Levels (ng/mL) | baseline and 12 weeks
  The levels of leptin will be determined by enzyme immunoassay (SPI BIO, Montigny le Bretonneux, France) using a plate reader (Biochrom Anthos MultiRead 400, Biochrom Ltd., Cambridge, UK).
Body Fat Percentage (%) | baseline and 12 weeks
  The body fat percentage will be determined measuring the skinfolds at seven sites (triceps, subscapular, suprailiac, axillary, pectoral, abdomen and thigh) using a standardized technique of measurement and determination.
Number of Oocytes Retrieved | between 12 and 16 weeks, during the in vitro fertilization cycle
  Women will follow a pre-established protocol of ovarian stimulation as part of the preparation for the in vitro fertilization cycle. The evolution of oocytes development will be accompanied by the medical team using the ultrasound technique and when at least one oocyte reach the average size of 17 mm the puncture of oocytes by aspiration will be held.
Percentage of Fertilized Oocytes (%) | between 12 and 16 weeks, during the in vitro fertilization cycle
  The percentage of fertilized oocytes will be obtained using the following formula: number of embryos/ total number of oocytes x 100.
Embryo Quality | between 12 and 16 weeks, during the in vitro fertilization cycle
  Embryo quality will be determined by the Embryonic Score Calculation - ESC, where embryos with score 4, are considered the best quality.

CONTACTS AND LOCATIONS:
Overall Officials: Cileide C Moulin, PhD, Principal Investigator — UFRGS/HCPA
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Cummings DE, Foster-Schubert KE, Overduin J. Ghrelin and energy balance: focus on current controversies. Curr Drug Targets. 2005 Mar;6(2):153-69. doi: 10.2174/1389450053174569. PMID 15777186
- [Background] Jackson AS, Pollock ML. Generalized equations for predicting body density of men. Br J Nutr. 1978 Nov;40(3):497-504. doi: 10.1079/bjn19780152. PMID 718832
- [Background] Loret de Mola JR. Obesity and its relationship to infertility in men and women. Obstet Gynecol Clin North Am. 2009 Jun;36(2):333-46, ix. doi: 10.1016/j.ogc.2009.03.002. PMID 19501317
- [Background] Marfell-Jones, M., Olds, T., Stewart, A., and Carter, J.E.L. 2006. International standards for anthropometric assessment. North-West University, Potchefstroom, RSA.
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Metwally M, Ledger WL, Li TC. Reproductive endocrinology and clinical aspects of obesity in women. Ann N Y Acad Sci. 2008 Apr;1127:140-6. doi: 10.1196/annals.1434.000. PMID 18443342
- [Background] Singla P, Bardoloi A, Parkash AA. Metabolic effects of obesity: A review. World J Diabetes. 2010 Jul 15;1(3):76-88. doi: 10.4239/wjd.v1.i3.76. PMID 21537431
- [Background] Sliwowska JH, Fergani C, Gawalek M, Skowronska B, Fichna P, Lehman MN. Insulin: its role in the central control of reproduction. Physiol Behav. 2014 Jun 22;133:197-206. doi: 10.1016/j.physbeh.2014.05.021. Epub 2014 May 27. PMID 24874777
- [Background] Terriou P, Sapin C, Giorgetti C, Hans E, Spach JL, Roulier R. Embryo score is a better predictor of pregnancy than the number of transferred embryos or female age. Fertil Steril. 2001 Mar;75(3):525-31. doi: 10.1016/s0015-0282(00)01741-6. PMID 11239536
- [Background] Zegers-Hochschild F, Adamson GD, de Mouzon J, Ishihara O, Mansour R, Nygren K, Sullivan E, Vanderpoel S; International Committee for Monitoring Assisted Reproductive Technology; World Health Organization. International Committee for Monitoring Assisted Reproductive Technology (ICMART) and the World Health Organization (WHO) revised glossary of ART terminology, 2009. Fertil Steril. 2009 Nov;92(5):1520-4. doi: 10.1016/j.fertnstert.2009.09.009. Epub 2009 Oct 14. PMID 19828144
- [Derived] Becker GF, Passos EP, Moulin CC. Short-term effects of a hypocaloric diet with low glycemic index and low glycemic load on body adiposity, metabolic variables, ghrelin, leptin, and pregnancy rate in overweight and obese infertile women: a randomized controlled trial. Am J Clin Nutr. 2015 Dec;102(6):1365-72. doi: 10.3945/ajcn.115.117200. Epub 2015 Nov 11. PMID 26561614